CLINICAL TRIAL: NCT04540328
Title: Effect of Non-surgical Peridontal Treatment on Cardiovascular Risk Markers in Patients With Severe Chronic Periodontitis
Brief Title: Non-surgical Peridontal Treatment on Cardiovascular Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Assistant Professor, Kırıkkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015 / 029
Record Dates: First submitted 2018-03-07; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Risk Markers; Chronic Periodontitis
Keywords: asymmetric dimethylarginine; endothelial nitric oxide synthase; homocysteine; monocyte chemoattractant protein-1
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-surgical peridontal treatment (Other): Patients with chronic periodontitis received non-surgical periodontal treatment, including scaling and root planing and polishing within 14 days under local anesthesia with manual and ultrasonic devices and standardized oral hygiene instructions including methods of tooth-brushing and interdental cleaning were also given to each one. A professional supragingival plaque control was applied on a regular basis every month.
  Interventions: Other: Non-surgical periodontal treatment

INTERVENTIONS:
Other: Non-surgical periodontal treatment

SUMMARY:
The study evaluates the influence of non-surgical mechanical periodontal treatment in patients with severe chronic periodontitis on inflammatory markers related to risk for cardiovascular diseases

DETAILED DESCRIPTION:
A total of 80 non-smokers with systemically healthy, including 40 patients with severe chronic periodontitis and 40 periodontally health subjects were included into the present study. The probing depth, clinical attachment level, plaque index, gingival index and blood samples were collected at baseline and at the 3rd months after treatment and the serum levels of asymmetric dimethylarginine (ADMA), endothelial nitric oxide synthase (eNOS), homocysteine (Hcy), monocyte chemoattractant protein-1 (MCP-1) were determined with enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of severe chronic periodontitis

Clinical diagnosis of periodontal health

Exclusion Criteria:

Systemic diseases such as diabetes, cardiovascular disease

Periodontal treatment within the previous year

Drugs such as systemic steroids, non-steroidal anti-inflammatory drugs, immunosuppressants, hormone drugs, contraceptives, anticoagulants, cholesterol regulating drugs, systemic antibiotics, antioxidants within the previous 3 months

Pregnant or lactating

Consumed alcohol

Smoker

Ages: 30 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Asymmetric dimethylarginine (ADMA) | At the 3rd months after non-surgical periodontal treatment
  Serum Concentration (pg/mL)
Endothelial nitric oxide synthase (eNOS) | At the 3rd months after non-surgical periodontal treatment
  Serum Concentration (pg/mL)
Homocysteine (Hcy) | At the 3rd months after non-surgical periodontal treatment
  Serum Concentration (nmol/mL)
Monocyte chemoattractant protein-1 (MCP-1) | At the 3rd months after non-surgical periodontal treatment
  Serum Concentration (ng/mL)

SECONDARY OUTCOMES:
Clinical periodontal parameter | At the 3rd months after non-surgical periodontal treatment
  Clinical attachment level (mm)